CLINICAL TRIAL: NCT05159674
Title: Study on the Difference and Cause of Acupuncture Dexmedetomidine Compound Anesthesia Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021.11.30
Record Dates: First submitted 2021-11-30; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Acupuncture; Dexmedetomidine; Anesthesia
Keywords: Acupuncture; Dexmedetomidine; Combined anesthesia; Metabolic enzyme

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine+electroacupuncture compound anesthesia (Experimental): EA was given every day three days before surgery, 30 minutes before induction of anesthesia + the whole course of surgery, and every 12 hours from the first day after surgery, each treatment was performed for 30 minutes until 48 hours after surgery. During the operation, only dexmedetomidine was used to make BIS<80.
  Interventions: Device: Dexmedetomidine+electroacupuncture compound anesthesia
- Dexmedetomidine anesthesia (No Intervention): There was no EA treatment before, during or after operation. During the operation, only dexmedetomidine was used to make BIS<80.

INTERVENTIONS:
Device: Dexmedetomidine+electroacupuncture compound anesthesia — Dexmedetomidine and acupuncture were given together to induce anesthesia
  Arms: Dexmedetomidine+electroacupuncture compound anesthesia

SUMMARY:
Studies have shown that the use of dexmedetomidine before and during surgery has a good sedative, analgesic and circulatory stabilizing effect. The use of dexmedetomidine in thoracoscopic lung resection has been proven to be safe and feasible, and it has a certain degree of improvement in postoperative lung function. Combining the advantages of thoracoscopy and the previous experience of combined acupuncture and drug anesthesia technology, our team pioneered cardiopulmonary surgery without endotracheal intubation and combined needle and drug anesthesia, so that the patient was in a state of light sleep and spontaneous breathing without tracheal intubation. After completing the operation, it was found that this technical method can effectively reduce the amount of intraoperative anesthetics, improve intraoperative lung ventilation, improve lung oxygenation, achieve intraoperative organ protection, and significantly reduce complications caused by tracheal intubation , Postoperative analgesic drugs have reduced the amount of 20%, accelerate the time of exhaust and defecation, and its postoperative rehabilitation is better than conventional treatment. These results suggest that the combination of acupuncture and medicine is not only suitable for anesthesia, it can be used scientifically and rationally in postoperative analgesia, immune regulation and even the entire perioperative organ protection, creating more possibilities for patients' ERAS.

In combined acupuncture and drug anesthesia, the core goal is to use acupuncture to reduce the insufficiency of anesthetics in terms of analgesia, sedation, stable circulation, and protection of organs. However, the mechanism of action behind this type of combination has not yet been improved. Efficacy kinetics or pharmacokinetics has been explained convincingly, or it is not well recognized. For example, is there a specific target in the body of acupuncture? If there is a specific target, where is the effect target? If the combined application of acupuncture and medicine produces a synergistic effect through a pharmacokinetic mechanism, its specific mechanism still needs to be clarified.

DETAILED DESCRIPTION:
Usually in a disease state, the body is in a state of strong stress, and the body's redox balance is disrupted. This state will also affect the activity of metabolic enzymes in the body, which in turn will have a corresponding impact on drug metabolism. Therefore, the body's basic redox level The monitoring of the drug is very important for the clinical development of individualized dosing regimens and the combined acupuncture and drug anesthesia mechanism.

Modern pharmacokinetic studies have shown that 90% of drugs (including most anesthetics) will undergo the metabolism of CYP enzyme and UGT enzyme, that is, their substrates. These drugs are mostly used in combination of multiple drugs in clinical practice. Therefore, it is not only necessary to study the individual change law of its single drug use, but also the change law of its multi-drug sharing and mutual influence. The original intention of sharing or combining drugs is to be beneficial to the patient, but when the common interaction between the shared drug and the original drug has a harmful effect on the body, adverse drug reactions will occur, which is also called drug-drug interaction (Drug-Drug Interaction DDI), and the production of DDI is nothing more than pharmacodynamics or pharmacokinetic interactions. Therefore, when combining drugs or combined acupuncture and drug anesthesia, it is also necessary to monitor the effects and effects of metabolic enzymes in the body on the drugs first, and then to determine the safety and the mechanism of the effect of multi-drug sharing.

It has been reported that the combination of acupuncture and medicine produces pharmacodynamic effects such as increased endorphins, reduction of stress, immune function regulation, and up-regulation of endorphin receptor activity. Therefore, this study will start from these aspects. To design research on the mechanism of combined acupuncture and drug anesthesia, we hope to observe objective evidence of pharmacokinetics or pharmacodynamics that significantly reduces the use of anesthetics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pulmonary nodules scheduled for thoracoscopic surgery;
2. Age ≥ 18 and ≤ 75, regardless of gender;
3. Understand and agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Patients who have previously received EA treatment;
2. Patients with skin infection at acupoints;
3. Patients with nerve injury of upper or lower limbs;
4. Those who have participated or are participating in other clinical trials one month before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Time required for bispectral index of EEG to be less than 80 | From the time anesthesia was given until the end time of the surgery
  The time required for bispectral index of EEG in the intervention group was lower than that in the non intervention group